CLINICAL TRIAL: NCT06390891
Title: Importance of Patient Characteristics in Identifying and Selecting Patients Suitable for Pancreatic Resection
Brief Title: Role of Patient Selection for Pancreatic Resections
Acronym: PatSelPanc
Status: Completed | Type: Observational
Sponsor: Medizinische Hochschule Brandenburg Theodor Fontane (Other)
Responsible Party: Principal Investigator, Rene Mantke, Head of Surgery, Medizinische Hochschule Brandenburg Theodor Fontane
Other Study IDs: PatSelPanc
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Pancreas Disease
Keywords: Specialization; Pancreatic Surgery; Resection; Volume-Outcome-Relationship
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients treated in high-volume pancreatic centers: Patients treated at a hospital performing at least 50 pancreatic resection procedures annually during 2010 to 2018
  Interventions: Other: Persons with pancreatic resection in a hospital with at least 50 pancreatic resections annually (observational),
- Patients treated in low-volume pancreatic centers: Patients not treated at a hospital performing at least 50 pancreatic resection procedures annually during 2010 to 2018
  Interventions: Other: Persons with pancreatic resection in a hospital not performing at least 50 pancreatic resections annually (observational),

INTERVENTIONS:
Other: Persons with pancreatic resection in a hospital with at least 50 pancreatic resections annually (observational), — Persons that have undergone a pancreatic resection at a hospital with at least 50 pancreatic resections annually (observational)
  Groups: Patients treated in high-volume pancreatic centers
Other: Persons with pancreatic resection in a hospital not performing at least 50 pancreatic resections annually (observational), — Persons that have undergone a pancreatic resection at a hospital with not at least 50 pancreatic resections annually (observational)
  Groups: Patients treated in low-volume pancreatic centers

SUMMARY:
Pancreatic surgery is complicated and risky, especially for pancreatic cancer. It's been noticed that having these surgeries done at specialized centers can lead to better outcomes and survival rates. However, factors like patient selection and hospital conditions also play an important role. Some studies show that more surgeries done at a hospital might not always mean better results, as the type of patients and procedures can vary. To understand this better, the present study compared outcomes and patient characteristics between high-volume pancreatic centers and others.

DETAILED DESCRIPTION:
The study utilized German nationwide administrative data (diagnosis-related group statistics) spanning from 2010 to 2018. Persons who underwent pancreatic resections during this period were included, with exclusions for certain criteria like underage and type of procedure. Various factors including patient demographics, diagnoses, procedures, and comorbidities were analyzed to assess in-hospital mortality rates. High-volume pancreatic centers (HVPCs) were identified as those performing at least 50 procedures annually. Statistical analyses included comparing crude and adjusted mortality rates and assessing patient characteristics between HVPCs and non-HVPCs. Models were adjusted for multiple variables, and methods like the Cochran-Armitage trend test and mixed models were employed. Additionally, the study investigated how differences in patient characteristics between HVPCs and non-HVPCs affected mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* partial or total pancreatic resections between 2010 and 2018

Exclusion Criteria:

* childhood (<18 years)
* subjects with a pancreatic transplantation procedure
* missing information on age or gender

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population encompasses all patients that underwent any pancreatic resection procedure in any German hospital (full survey of the German population).
Sampling Method: Non-Probability Sample
Enrollment: 86073 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | 30 days
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Rene Mantke, MD, PhD, Study Director — Head of Surgery at University Hospital Brandenburg an der Havel

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not available for data sharing.

REFERENCES:
- [Derived] Mantke R, Seliger B, Ogino S, Buchler MW, Hunger R. Not Only Caseload but Also Patient Selection Is Predictive of Mortality After Pancreatic Resection. Ann Surg Open. 2024 Dec 30;6(1):e536. doi: 10.1097/AS9.0000000000000536. eCollection 2025 Mar. PMID 40134472